CLINICAL TRIAL: NCT00164970
Title: Can Oral Vitamin B12 and Folate Supplementation Preserve Cognitive Function of Patients With Early Dementia?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT-B12
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Vitamin B 12; Folic Acid

INTERVENTIONS:
Dietary Supplement: Vitamin B12
Dietary Supplement: folate

SUMMARY:
Background: Vitamin B12 and folate are essential to brain health. Sub optimal status of vitamin B12 and folate leads to elevation of plasma homocysteine concentration, which is associated with Dementia. Vitamin B12 and folate supplementation improved the cognitive function of demented subjects with hyperhomocysteinaemia in a pilot study.

Objective: To determine the effectiveness of vitamin B12 and folate supplementation in preserving cognitive function of subjects with early dementia

DETAILED DESCRIPTION:
After stratified randomization by mini mental state examination scores, supplement group subjects take 1 mg of methylcobalamin and 5 mg of folic acid daily, while placebo group subjects take placebo capsules. The primary outcome is Mattis dementia rating scale. The secondary outcomes are mini mental state examination, neuropsychiatric inventory, and Cornell scale for depression in dementia. These measurements will be performed at baseline and every six months for 24 months. Fasting plasma homocysteine concentrations are measured at baseline and 18-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Dementia of Alzheimer's or vascular type
* Early dementia defined by Clinical Dementia Rating of 1.

Exclusion Criteria:

* lives alone
* significant communication problems
* significant co-existing diseases
* blood tests:vitamin B12< 150 pmol/l, serum creatinine> 250 mol/l, hypothyroidism and syphilis

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2004-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
dementia rating scale | at 6 months, 12 months and 18 months
depression rating scale | at 6 months, 12 months and 18 months

SECONDARY OUTCOMES:
vitamin b12 | at 18 months
folate | at 18 months
homocysteine | at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy CY Kwok, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong, China